CLINICAL TRIAL: NCT03265717
Title: A Phase II Study of INVAC-1 as Treatment of Patients With High-risk Chronic Lymphocytic Leukemia
Brief Title: DNA Plasmid Encoding a Modified Human Telomerase Reverse Transcriptase (hTERT), Invac-1 in Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor decision
Sponsor: Invectys (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INVAC1-CT-201
Record Dates: First submitted 2017-08-24; First posted 2017-08-29 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
Keywords: telomerase, tert, cancer vaccine
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Untreated high risk "watch and wait" (Experimental): Newly diagnosed patients not eligible for any approved treatment (using NCI Working Group criteria), but having some poor prognosis characteristics (defined by MDACC nomogram criteria). Patients will be treated by INVAC-1 for 6 months and then MRD will be assessed. Patients will subsequently be managed as per usual care. For MRD negative patients after INVAC-1 who become MRD+ during follow-up, INVAC-1 can be resumed for one year.
  Interventions: Biological: INVAC-1
- Group 2: Ibrutinib treated patients (Experimental): Patients who are receiving ibrutinib as 1st or 2nd line treatment. After at least 12 months of ibrutinib, patients will be assessed for MRD. MRD-positive patients will be treated with ibrutinib + INVAC-1 for 6 months and at the end of the combined treatment period, MRD will be assessed. MRD-negative patients (defined as <0.01% of CLL cells in total cells analyzed) will have the option to stop or continue ibrutinib. Then, they will be followed-up regularly for two years. Patients who become MRD-positive after being MRD-negative will resume ibrutinib single agent.
  Interventions: Biological: INVAC-1

INTERVENTIONS:
Biological: INVAC-1 — Patients are treated by INVAC-1 for 6 cycles at 4-week intervals

SUMMARY:
Phase 2 study to assess the efficacy of INVAC-1, a DNA plasmid encoding a modified human telomerase reverse transcriptas (hTERT) protein, at a dose of 800 µg for 6 cycles 4 weeks apart on Minimal Residual Disease (MRD) eradication rate in the bone marrow, either as a single agent in a high risk "watch and wait" group (group 1 - 42 patients) or in combination with ibrutinib (group 2 - 42 patients), in patients with Chronic Lymphocytic Leukemia (CLL).

Pharmacodynamics and safety will also be assessed.

DETAILED DESCRIPTION:
The study will be a phase II, open label, single-arm trial of INVAC-1 at a dose of 800 µg in patients with CLL.

The primary goal of the study is to achieve MRD negativity in each group. 42 patients are to be included in each study group.

Group 1: Untreated high risk "watch and wait" Newly diagnosed patients not eligible for any approved treatment (using NCI Working Group criteria), but having some poor prognosis characteristics (defined by MD Anderson Cancer Center nomogram criteria). Patients will be treated by INVAC-1 for 6 doses at 4-week intervals and then MRD will be assessed. Patients will subsequently be managed as per usual care. For MRD negative patients after INVAC-1 who become MRD+ during follow-up, INVAC-1 can be resumed for 6 months.

Group 2: Ibrutinib treated patients Patients who are receiving ibrutinib as 1st or 2nd line treatment. After at least 12 months of ibrutinib, patients will be assessed for MRD. MRD-positive patients will be treated with ibrutinib + INVAC-1 for 6 months and at the end of the combined treatment period, MRD will be assessed. MRD-negative patients (defined as <0.01% of CLL cells in total cells analyzed) will have the option to stop or continue ibrutinib. Then, they will be followed-up regularly for two years. Patients who become MRD-positive after being MRD-negative will resume ibrutinib single agent.

ELIGIBILITY:
Group 1: Untreated high risk "watch and wait"

Inclusion Criteria:

1. Age ≥ 18 years old
2. Rai stage 0 - II without active disease according to IWCLL 2018 criteria
3. Predicted time to first treatment of ≤3 years according to MDACC nomogram.
4. ECOG performance status of 0-2
5. Adequate hepatic function, defined as serum aspartate transaminase (AST) and alanine transaminase (ALT) < 2.5 x upper limit of normal (ULN), and total bilirubin ≤ 1.5 x ULN except Gilbert's Syndrome where a direct bilirubin ≤ 1.5 ULN will be used.
6. Adequate renal function, defined as an estimated creatinine clearance ≥30 mL/min using the Cockcroft-Gault equation
7. Willingness to receive all outpatient treatment, all laboratory monitoring, and all radiological evaluations at the institution that administers study drug for the entire study
8. Willingness of male and female patients, if sexually active, to use an effective barrier method of contraception during the study and for 3 months following the last dose of study drug
9. Ability to provide written informed consent and to understand and comply with the requirements of the study

Exclusion Criteria

1. Any investigational agent(s) within 4 weeks prior to entry
2. Uncontrolled autoimmune hemolytic anemia (Hgb < 11g/deciliter) or idiopathic thrombocytopenic purpura (< 100,000/µl)
3. Any previous treatment (chemotherapy, radiotherapy, and/or monoclonal antibodies) intended specifically to treat CLL
4. Treatment with corticosteroids other than physiological replacement within the previous week or treatment with immunosuppressive medication within the previous week.
5. Major surgery within 4 weeks prior to inclusion
6. Currently active, clinically significant cardiovascular disease or a history of myocardial infarction within 6 months prior to inclusion
7. Uncontrolled active systemic fungal, bacterial, viral, or other infection or requirement for intravenous (IV) antibiotics
8. Known history of infection with human immunodeficiency virus (HIV)
9. Serologic status reflecting active hepatitis B or C infection.
10. History of stroke or intracranial hemorrhage within 6 months prior to enrolment
11. Current life-threatening illness, medical condition, or organ-system dysfunction that could compromise patient safety or put the study at risk
12. Breast-feeding or pregnant women, or patients for whom there is a risk of conception and who are unable or unwilling to use appropriate contraception (for male and female patients up to 4 months after end of ibrutinib.)
13. Previous malignancy with life expectancy less than 6 months or requiring systemic treatment (except colorectal cancer, history of basal cell carcinoma of skin or pre-invasive carcinoma of the cervix with adequate treatment)
14. Known drug abuse/ alcohol abuse
15. Severe organ failures or diseases, including: clinically relevant coronary disease, myocardial infarction or any other relevant cardiovascular disorder within 12 months before study entry, severe psychiatric illness and severe infection.

Group 2: Ibrutinib treated patients

Inclusion Criteria

1. Age ≥ 18 years old
2. Males or females with CLL diagnosed according to IWCLL diagnostic criteria who have been treated with ibrutinib therapy for at least 12 months and have had no more than 1 other treatment for CLL prior to receiving ibrutinib.
3. Currently in complete or partial remission (PR)/PR with lymphocytosis (PRL)
4. MRD positivity defined as >0.5% CLL cells in the bone marrow by flow cytometry
5. ECOG performance status of 0-2
6. Adequate hepatic function, defined as serum aspartate transaminase (AST) and alanine transaminase (ALT) < 2.5 x upper limit of normal (ULN), and total bilirubin ≤ 1.5 x ULN, unless Gilbert's Syndrome where a direct bilirubin ≤ 1.5 ULN will be used.
7. Adequate renal function, defined as estimated creatinine clearance ≥ 30 mL/min using the Cockcroft-Gault equation
8. Willingness to receive all outpatient treatment, all laboratory monitoring, and all radiological evaluations at the institution that administers study drug for the entire study
9. Willingness of male and female patients, if sexually active, to use an effective barrier method of contraception during the study and for 3 months following the last dose of study drug
10. Ability to provide written informed consent and to understand and comply with the requirements of the study

Exclusion Criteria

1. Any investigational agent(s) within 4 weeks prior to entry
2. Known involvement of the central nervous system by lymphoma or leukemia
3. History or current evidence of Richter's transformation or prolymphocytic leukemia
4. Uncontrolled autoimmune hemolytic anemia (Hgb < 11g/deciliter) or idiopathic thrombocytopenic purpura (< 100,000/µl)
5. More than one previous treatment by chemotherapy or patients who previously received alemtuzumab intended specifically to treat CLL
6. Corticosteroid use within 1 week prior to first dose of study drug, with the exception of inhaled, topical, or other local administrations. Patients requiring systemic steroids at daily doses > 20 mg prednisone (or corticosteroid equivalent), or those who are administered steroids for leukemia control or white blood cell (WBC)-count-lowering are excluded
7. Major surgery within 4 weeks prior to inclusion
8. Currently active, clinically significant cardiovascular disease or a history of myocardial infarction within 6 months prior to inclusion
9. Uncontrolled active systemic fungal, bacterial, viral, or other infection or requirement for intravenous (IV) antibiotics
10. Known history of infection with human immunodeficiency virus (HIV)
11. Serologic status reflecting active hepatitis B or C infection
12. History of stroke or intracranial hemorrhage within 6 months prior to enrollment
13. Current life-threatening illness, medical condition, or organ-system dysfunction that could compromise patient safety or put the study at risk
14. Requirement for anticoagulation with warfarin, or for treatment with a strong CYP3A4/5 and/or CYP2D6 inhibitor
15. Breast-feeding or pregnant women, or patients for whom there is a risk of conception and who are unable or unwilling to use appropriate contraception (for male and female patients up to 4 months after end of ibrutinib.)
16. Previous malignancy with life expectancy less than 6 months or requiring systemic treatment (except colorectal cancer, history of basal cell or squamous carcinoma of skin or pre-invasive carcinoma of the cervix with adequate treatment)
17. Known drug abuse/ alcohol abuse
18. Severe organ failures or diseases, including: clinically relevant coronary disease, myocardial infarction or any other relevant cardiovascular disorder within 12 months before study entry, severe psychiatric illness and severe infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Minimal Residual Disease (MRD) eradication rate in the bone marrow | 6 months
  MRD eradication rate (by standardized 4-color flow cytometry, with a limit of detection of 0.01% CLL cells among total leucocytes in the bone marrow after 6 monthly injections of INVAC-1

SECONDARY OUTCOMES:
MRD eradication rate in blood after 6 monthly injections of INVAC-1 | 6 months
Duration of MRD eradication in bone marrow and blood | approximately 3 years
Cumulative incidence of partial and complete response by IWCLL 2018 | every 6 months for 3 years
PFS as assessed by investigators according to IWCLL 2018 criteria | approximately 3 years
Time to next CLL treatment | approximately 3 years
Overall survival | approximately 3 years
Adverse events | up to 7 months
  type, frequency, severity as graded by NCI CTCAE v.4.03
Cellular (CD4 & CD8) specific anti hTert response by FACS including cytokine polarization Th1, Th2, Th17 | every 6 months for 3 years
Count of blood circulating CD4, CD8, Treg, NK cells | every 6 months for 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided